CLINICAL TRIAL: NCT00389012
Title: Strength Training Effectiveness Post-Stroke (STEPS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Physical Therapy Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 025024
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2010-04

CONDITIONS: Cerebrovascular Accident
Keywords: rehabilitation; hemiplegic gait; exercise therapy; physical therapy
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Exercise Therapy

INTERVENTIONS:
Procedure: exercise therapy
Procedure: walking rehabilitation

SUMMARY:
The purpose of this study is to determine if treadmill training with body weight-support (BWST) is more effective at improving walking in individuals post-stroke than a resisted leg-cycling exercise program. In addition, we want to determine if training programs that combine leg strength training to treadmill walking provide an additional benefit to post-stroke walking outcomes.

DETAILED DESCRIPTION:
Impaired walking ability is a hallmark residual deficit that contributes to post-stroke walking disability . Impairment in lower extremity muscle strength is a significant contributor to decreased walking speed after stroke. No studies have combined task-specific locomotor training in combination with lower extremity strength training programs designed to improve post-stroke walking outcomes.

Participants will include individuals who are ambulatory, but walk slower than 1.0 m/sec and are at least 6 months post unilateral stroke.

Participants are stratified by initial comfortable walking speed (moderate >0.5 m/sec; severe <= 0.5 m/sec) and randomized to one of four exercise pairs: 1) body-weight supported treadmill training (BWST) and locomotor-based strength training (resistive cycling task, LBST), 2) BWST and LE muscle-specific strength training (MSST), 3) BWST and upper extremity ergometry (SHAM), and 4) LBST and SHAM. Training will occur 4 times per week for 6 weeks (24 total sessions). Exercise type in each exercise pair is alternated daily.

Primary outcomes include comfortable and fast overground walking speed, and distance walked in 6-minutes measured at baseline, after 12 and 24 treatment sessions and at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* 4 months to 5 years after first-time onset of a ischemic or hemorrhagic cerebrovascular accident (CVA) confirmed by CT, MRI, or clinical criteria
* able to ambulate at least 14 meters with assistive and/or orthotic device and one person assist (minimum Functional Ambulation Classification Level II
* self-selected walking velocity of ≤1.0 meters/second
* approval of primary care physician to participate.

Exclusion Criteria:

* resting systolic blood pressure greater than 180mmHg and/or diastolic blood pressure greater than 110mmHg and/or resting heart rate greater than 100 beats/minute;
* lower limb orthopedic conditions such as prior joint replacement or range of motion limitations;
* spasticity management that included Botox injection (< 4 months earlier) or phenol block injection (< 12 months earlier) to affected lower extremity and intrathecal Baclofen or oral Baclofen (within past 30 days);
* Mini-Mental State Exam score < 24;
* currently receiving lower extremity strengthening exercises or gait training,
* past participation in any study examining the effects of long term (>4 weeks training) body weight support treadmill training; limb loaded pedaling, or lower extremity strengthening;
* plans to move out of the area in the next year,
* no transportation to the study site for all evaluations and intervention sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-05; Primary Completion 2010-10-31 (Actual); Study Completion 2010-10-31 (Actual)

PRIMARY OUTCOMES:
walking speed (meters/second)
walking distance (distance walked in 6-minutes)

SECONDARY OUTCOMES:
Lower extremity Fugl-Meyer
Berg Balance Score
Lower extremity torque
Stroke Impact Scale
SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Katherine J Sullivan, PhD, PT, Principal Investigator — Division of Biokinesiology and Physical Therapy, University of Southern California, Los Angeles, California; David A Brown, PhD, PT, Principal Investigator — Department of Physical Therapy and Movement Sciences, Feinberg School of Medicine, Northwestern University, Chicago, Illinois; Sara Mulroy, PhD, PT, Principal Investigator — Pathokinesiology Laboratory, Rancho Los Amigos National Rehabilitation Center, Downey, California
Locations (3):
- United States (3):
  - Rancho Los Amigos, Downey, California
  - University of Southern California, Los Angeles, California
  - Northwestern University, Chicago, Illinois

REFERENCES:
- [Derived] Sullivan KJ, Brown DA, Klassen T, Mulroy S, Ge T, Azen SP, Winstein CJ; Physical Therapy Clinical Research Network (PTClinResNet). Effects of task-specific locomotor and strength training in adults who were ambulatory after stroke: results of the STEPS randomized clinical trial. Phys Ther. 2007 Dec;87(12):1580-602. doi: 10.2522/ptj.20060310. Epub 2007 Sep 25. PMID 17895349